CLINICAL TRIAL: NCT01663779
Title: Comparison of Ultrasound-guided Versus Blind Insertion of Radial Artery Catheters.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit further.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1206010421
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound radial artery catheter (Experimental): Ultrasound guided radial artery catheterization.
  Interventions: Procedure: Ultrasound guided radial artery catheterization.
- Palpation based artery catheterization (Active Comparator): Blind insertion of radial artery catheterization
  Interventions: Procedure: Blind insertion of radial artery catheterization

INTERVENTIONS:
Procedure: Ultrasound guided radial artery catheterization. — Radial artery catheters will be placed with the assistance of bedside ultrasound.
  Arms: Ultrasound radial artery catheter
Procedure: Blind insertion of radial artery catheterization — Radial artery catheters will be placed by the palpation technique only.
  Arms: Palpation based artery catheterization

SUMMARY:
Arterial catheterization is frequently performed on critically ill patients for invasive blood pressure monitoring and/or frequent blood draws, especially arterial blood gas analysis. The distal part of the radial artery (wrist) is the preferred access site.

The potential complications of the procedure are mostly minor and comprise temporary occlusion of the radial artery (RA), hematoma, local infection or bleeding from the puncture site. Major complications including vessel aneurysm or occlusion with threat to hand viability are rare.

The standard approach to catheterization is "blind" puncture of the RA while locating its pulse by palpation, followed by threading a 20 Gauge (20G) angio-catheter into the vessel. Alternatively ultrasound can be used to locate the vessel and guide needle insertion.

To our knowledge, four prospective randomized trials (PRT)5-8 comparing palpation with ultrasound-guided RA catheterization have been conducted so far and one meta-analysis looked at the pooled data obtained from these. The results showed that ultrasound guidance increased the first-attempt success rate at RA catheterization by 71% compared to palpation. The use of ultrasound also significantly reduced the time to successful catheterization, the number of punctures as well as the amount of catheters required per procedure.

None of the prior randomized trials has been conducted in an ICU setting and in three out of the four studies the arterial lines were placed in patients undergoing elective surgery. The investigators hypothesized that ultrasound could improve first attempt success rate while placing arterial catheters in an ICU setting. Ultrasound may also reduce total time to successful insertion and reduce complications.

The investigators plan to randomize patients to either a palpation technique or ultrasound guided catheter insertion and record the above outcomes.

DETAILED DESCRIPTION:
The study will be conducted in a prospective randomized design on the patient population of the Surgical Intensive Care Unit (SICU) at Yale New Haven Hospital. All SICU patients in whom the indication for arterial catheterization has been established by the attending physician will be eligible for consented randomization to either the "Palpation" or the "Ultrasound" group.

Once consent from the patient or his/her surrogate has been obtained, eligible patients will be randomized to either the "Palpation" or the "Ultrasound" group. Sequentially numbered sealed envelopes will be maintained in the SICU.

Catheter insertion: The side of insertion (left/right arm) is chosen by the operator. The wrist is positioned by the operator, the skin disinfected and the area draped in a sterile fashion. "Palpation" group": The artery is punctured after location by palpation only. "Ultrasound" group": The artery is punctured under real-time ultrasound only with the probe draped in a sterile sheath. The time from the first skin puncture to confirmed intra-arterial position of the catheter by observing blood return from the catheter is measured with a chronometer by a second person. An arterial pressure waveform must be observed on the monitor to validate intra-arterial catheter placement.

Radial artery cannulation will be performed using the "Radial Artery Catheterization Set with Integral Needle Protection" (Ref. RA-04020-SP, Arrows International Inc., Reading PA 19605, USA) containing a 20G catheter on a 22 gauge (22G) puncture needle and a 0.46 mm spring-wire guide.

For ultrasound-guided catheter insertion, operators will use the "Site-Rite 6 Ultrasound System" with a linear vascular access probe (5-10 MHz) (Bard Access Systems Inc., 605 North 5600 West, Salt Lake City, UT 84116, USA).

Operators: RA catheterization is a typical teaching procedure frequently performed in the ICU. In our unit, arterial lines are placed by either post graduate year 2 (PGY-2) residents (surgery & anesthesia) rotating through the SICU on a monthly basis, or by mid-level providers who are in the unit for indeterminate periods of time. For our study, this will be an important point, as one of our goals will be to demonstrate a learning effect, which is less likely to be observable among the PGY-2 residents who will be present in the unit for a month only.

All operators will get instructions (lecture and hands-on training on vascular phantom at the beginning of their SICU rotation) on the use of ultrasound for vascular access and will at all times have the opportunity to exercise their skills on a vessel phantom. Each successful vessel puncture on the vessel phantom must be recorded by the operator, including time and date. For each operator performing the ultrasound-guided insertion on a patient, one of the investigators will be present for supervision and data collection, but not for assistance with insertion, unless required for failure after having used both methods.

Cross-over: After three failed attempts at catheterization with the allocated first method, the alternative method must be used; the operator can opt to puncture the RA on the opposite arm. Timing of the first method ends when the operator decides to abandon the third attempt. Timing for the new method starts at the new first skin puncture.

Follow up: All catheters will be monitored daily and on days 1 and 3 with clinical and ultrasound examination for the development of complications. The catheter will be followed daily for functional outcomes defined as the quality of the arterial waveform on the monitor and the ability to draw blood from the catheter. The day on which the catheter ceases to function for each of these purposes will be recorded as well as the day of catheter removal.

ELIGIBILITY:
Inclusion Criteria:

* All surgical intensive care unit patients at Yale New Haven Hospital in whom the indication for arterial catheterization has been established by the attending physician will be eligible for consented randomization to either the "Palpation" or the "Ultrasound" group.

Exclusion Criteria:

* The patient or his/her surrogate declines to participate or the patient lacks a radial artery into which a catheter can be place.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Schuster, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound Radial Artery Catheter | Palpation Based Artery Catheterization
Started | 27 | 23
Completed | 27 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound Radial Artery Catheter | Palpation Based Artery Catheterization | Total
Number analyzed (Participants) | 27 | 23 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 18 | 40
  >=65 years | 5 | 5 | 10
Sex/Gender, Customized [Number; unit: participants] — Gender was not collected as a baseline variable.
  participants
    unknown | 27 | 23 | 50
Region of Enrollment [Number; unit: participants]
  United States | 27 | 23 | 50

OUTCOME MEASURES:

1. Primary Outcome: First Pass Success When Attempting Arterial Catheterization.
Description: first pass success when attempting arterial catheterization of the artery
Time Frame: Immediate, upon study entry
Measure: Number; unit: participants
Groups:
- Ultrasound: ultrasound atery
- Palpation: palpation artery
Arm/Group | Ultrasound | Palpation
Number analyzed (Participants) | 27 | 23
participants | 22 | 10
Statistical Analysis 1: Comparison: Ultrasound; Test type: Superiority or Other; p < 0.01, Chi-squared; Odds Ratio (OR) = 5, 95% CI 2-sided [3 to 7]

ADVERSE EVENTS:
Time Frame: entire study
Groups:
- Ultrasound: ultrasound artery
Arm/Group | Ultrasound | Palpation
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/23
Other Adverse Events (participants affected / at risk) | 1/27 | 0/23
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasound (N=27) | Palpation (N=23)
subcutaneous hematoma <1cm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — subcutaneous hematoma <1cm developed in 1 patient in the ultrasound group. Resolved with no intervention in 3 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No